CLINICAL TRIAL: NCT04451369
Title: Multicenter Randomized Study Comparing Neo Adjuvant Chemotherapy for Patients Managed for Ovarian Cancer With or Without a Connected Prehabilitation Program
Brief Title: Connected Prehabilitation Program During Neo Adjuvant Chemotherapy
Acronym: TRAINING
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Paoli-Calmettes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: TRAINING-01-IPC 2018-039
Record Dates: First submitted 2020-06-03; First posted 2020-06-30 (Actual); Last update posted 2021-02-10 (Actual); Status verified 2020-05

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): Group without prehabilitation program before surgery
- Prehabilitation group (Experimental): Group will follows a prehabilitation program before surgery
  Interventions: Other: Prehabilitation program

INTERVENTIONS:
Other: Prehabilitation program — physical, nutritional and psycho-social supports before surgery
  Arms: Prehabilitation group

SUMMARY:
NACT is a heavy oncologic treatment, which can impair functional capacity, nutritional and emotional status. These three impairments are often ignored and not taken into account in the pre-therapeutic evaluations but are correlated with postoperative morbidity and mortality after major surgery.

Recently, a prehabilitation before surgery, including physical, nutritional and psycho-social support, has been defined. From a literature review, the maximum oxygen uptake (VO2 max) seems to constitute a strong evaluation factor reflecting physical fitness, easily measured with a cardiopulmonary exercise test (CPET) at maximal effort.

Several studies have shown beneficial effects of trimodal prehabilitation programs on postoperative functional capacity, return to daily activities and pain relief.

Home-based program and connected devices may improve the feasibility and the compliance to this program.

The hypothesis of this study is that performing a connected supervised home-based and patient-tailored multimodal prehabilitation program from diagnosis to surgery (with or without ERAS program) during NACRT, for patients managed for ovarian cancer, will limit physical fitness alteration and will positively affect postoperative outcomes.

Our study consists in an early and multidimensional (combining nutritional, physical, emotional and medical support) prehabilitation program during NACT for patients with ovarian cancer, in order to limit physical alteration before surgical treatment, and therefore improve postoperative outcomes. It will include a home-based prehabilitation program, in order to allow care access to all eligible patients.

DETAILED DESCRIPTION:
The main objective will be to determine if a prehabilitation program during NACT, for patients treated for an advanced ovarian cancer will limit physical alteration before major abdomino-pelvic surgery, compared to a control group without prehabilitation program. The primary endpoint will be the comparison of the variation of VO2 max, between baseline and surgery, in the prehabilitation group vs control group: VO2 max will be measured with a cardiopulmonary exercise test (CPET) at maximal effort.

This prospective, multicentric randomized control trial will be conducted in 7 French comprehensive cancer Centers or University Hospital, in compliance with inclusion criteria. After an initial evaluation, patients will be randomized in two groups: Prehabilitation group (P group) and a Control group (C group).

For the P group, after baseline evaluation, we will be offering from diagnosis to surgery, during the NACT:

* A standardized, patient-tailored preoperative physical activity training program will be performed at home, from diagnosis to surgery. Supervision will be done with connected device (connected watches) and activity will be adapted,
* A nutritional care established in respect of the SFNEP-SFNCM guidelines. Nutritional support will be adapted by a dietician according to information transmitted daily (connected body fat weight scale),
* A psychological support with coping strategies.

For the C group: Patients with ovarian cancer will undergo NACT after baseline evaluation without prehabilitation program.

After NACT, for both groups, major abdomino-pelvic surgery will be done with or without ERAS pathway, according to the practice in each center.

ELIGIBILITY:
Inclusion Criteria:

1. Patient must have signed the written consent,
2. Age ≥ 18 years,
3. Patient with advanced ovarian cancer (AOC), FIGO Stage III - IV, undergoing surgery,
4. Patient with neo adjuvant chemotherapy (min 3 cycles, max 6 cycles),
5. Capability to perform a cardiopulmonary exercise test (CPET)
6. Patient affiliated to the national "Social Security" regimen or beneficiary of this regimen.

Exclusion Criteria:

1. Patient with cognitive impairment,
2. Pregnancy,
3. Neoadjuvant treatment contraindications,
4. Physical adapted activity program contraindication,
5. No possibility to have access to connected devices or do not have a smartphone or a computer
6. Patient deprived of liberty or placed under the authority of a tutor,
7. Patient considered socially or psychologically unable to comply with the procedure and the required medical follow-up.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Ovarian cancer.
Enrollment: 136 (Estimated)
Dates: Start 2021-05 (Estimated); Primary Completion 2022-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
To determine if a prehabilitation program during NACT, for patient managed with advanced ovarian cancer (AOC) will limit physical alteration before surgery, compared to a control group without prehabilitation program (change between 3 timepoints). | baseline, 15 days before surgery and 3 moths before surgery
  CHANGE of VO2 max between baseline (inclusion) and surgery (preoperative), in the prehabilitation group vs control group. VO2 max will be measured during a cardiopulmonary exercise test (CPET).

SECONDARY OUTCOMES:
to compare physical outcomes between both groups | baseline, before surgery, and 3 months after surgery
  o International Physical Activity Questionnaire (IPAQ) , administered at inclusion and at the time of surgery and after surgery
to compare physical outcomes between both groups | baseline, before surgery, and 3 months after surgery
  Muscular strength evaluated with dynamometer (brachial biceps)
to compare Quality of Life, emotional outcomes between both groups | baseline, before surgery, and 3 months after surgery
  Psychological status evaluated by the Hospital Anxiety and Depression Scale (HADS) (Annex 2)
to compare Quality of Life, emotional outcomes between both groups | baseline, before surgery, and 3 months after surgery
  Cancer related quality of life (QoL) evaluated by using the self-reported European Organization for Research and Treatment of Cancer (EORTC) core questionnaire (QLQ-C30) (Annex 3)
to compare Quality of Life, emotional outcomes between both groups | baseline, before surgery, and 3 months after surgery
  Motivation evaluated by a free interview and a coping strategy.
to compare nutritional outcomes between both groups | baseline, before surgery, and 3 months after surgery
  Change Body Mass Index (BMI)
to compare nutritional outcomes between both groups | baseline, before surgery, and 3 months after surgery
  Muscle mass evaluated with the Computed tomography-derived
to compare nutritional outcomes between both groups | baseline, before surgery, and 3 months after surgery
  skeletal muscle index measured by skeletal muscle mass cross-sectional area at L3/height2
to compare nutritional outcomes between both groups | baseline, before surgery, and 3 months after surgery
  Weight in kg
to compare Surgical Morbidity rate between both groups | at day 30 and day 90 (3 months) after surgery
  Clavien-Dindo classification
to compare Surgical Morbidity rate between both groups | at day 30 and day 90 (3 months) after surgery
  NCI-CTCAE v 5.0 classification

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lambaudie E, Bannier/Braticevic C, Villaron/Goetgheluck C, Zemmour C, Boher JM, Ben Soussan P, Pakradouni J, Brun C, Lopez Almeida L, Marino P. TRAINING-Ovary 01 (connecTed pRehabiliAtIoN pelvIc caNcer surGery): multicenter randomized study comparing neoadjuvant chemotherapy for patients managed for ovarian cancer with or without a connected pre-habilitation program. Int J Gynecol Cancer. 2021 Jun;31(6):920-924. doi: 10.1136/ijgc-2020-002128. Epub 2020 Dec 1. PMID 33262113